CLINICAL TRIAL: NCT00701740
Title: Phase II Randomized Controlled Trial to Evaluate the Clinical and Histological Effects of Oral Isotretinoin for the Treatment of Photoaging on Face and Forearms
Brief Title: Oral Isotretinoin for Photoaging: Results of a Randomized Controlled Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Edileia Bagatin, Edileia Bagatin, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIFESP
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Photoaging; Epidermal p53 Expression
Keywords: photoaging; isotretinoin; profilometry; digital analysis
MeSH Terms: interventions — Isotretinoin; terephthalylidene dicamphor sulfonic acid; drometrizole trisiloxane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): A - 21 subjects were treated 20mg isotretinoin 3/week plus moisturizer and sunscreen,for three months; 10 randomly selected were submitted to skin biopsies before and after the end of treatment
  Interventions: Drug: oral isotretinoin and Mexoryl SX / XL
- B (Active Comparator): 11 subjects received only the same moisturizer/sunscreen
  Interventions: Drug: Mexoryl XL / SX

INTERVENTIONS:
Drug: oral isotretinoin and Mexoryl SX / XL — 20mg, 3/week,continuously for three months
  Other Names: isotretinoin; mexoryl
  Arms: A
Drug: Mexoryl XL / SX — 11 subjects used only the same moisturizer and SPF 60 sunscreen
  Other Names: mexoryl
  Arms: B

SUMMARY:
A clinical and histological randomized controlled phase II trial to evaluate the efficacy and safety of oral isotretinoin for treating photoaging was performed with 32 menopausal or sterilized women aged 40-55y. The subjects were included in two randomly selected groups: A- 21 women received 20mg oral isotretinoin 3x week, moisturizer, sunscreen SPF 60 during three months; B- 11 women received only same moisturizer/sunscreen.

DETAILED DESCRIPTION:
Clinical assessment ranging from -2=very bad to +2=very good for all patients. Also, profilometry, corneometer and skin elasticity tests in periocular regions and left forearm; skin biopsy on left forearm before/after treatment in B and in 10 randomly selected patients from A. Microscopic evaluation of corneal layer and epidermal thickness, dermal elastosis, new collagen and p53 epidermal expression performed by quantitative digital image analysis. Blind evaluations (group/time) conducted by two independent observers.

Clinical evaluation results showed no alterations (0) or slight improvement (+1) for all patients; profilometry, corneometer and skin elasticity measurements presented a significant difference in pre and post treatment values (p=0,001 to 0,028) with no differences between A/B. Regarding histological findings and p53 expression no previous differences between groups before the treatment were observed (p>0,1).Quantitative microscopic digital analysis demonstrated no differences between groups at the end of the study for the majority of variables. However, slight but significant difference between A/B subjects was found for p53 with major expression reduction for those treated with oral isotretinoin [0,66±0,31 vs 0,94±0,34 respectively (p=0,04)]. The main side effects were cheilitis in 15 patients (75%) and xerophthalmia in 5 (25%). No significant alterations occurred in biochemical tests.

ELIGIBILITY:
Inclusion Criteria:

* menopausal or sterilized women

Exclusion Criteria:

* woman at risk of pregnancy, with alterations on liver function or lipid profile

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
histological findings | before and after 3 months

SECONDARY OUTCOMES:
laboratory tests | before, after 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edileia Bagatin, MD, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil